CLINICAL TRIAL: NCT01211223
Title: Effects of the Variation in the Time of Systemic Administration of Metronidazole and Amoxicillin Associated to the Non-surgical Therapy of Chronic Periodontitis.
Acronym: Metro + Amoxi
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Principal Investigator, Jorge Gamonal, Academic, University of Chile
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Facultad Odontologia, U Chile
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Periodontitis; Clinical and Microbiological Effects
Keywords: Chronic periodontitis; Metronidazole plus Amoxicillin; Mechanical periodontal therapy; Scaling and Root Planning; Periodontal treatment
MeSH Terms: conditions — Chronic Periodontitis | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Scaling and root planning + placebo + antibiotics (Experimental): * Scaling and root planning + placebo
  * Scaling and root planning + metronidazole plus amoxicillin
  * Metronidazole plus amoxicillin + scaling and root planning
  Interventions: Drug: Administration of Metronidazole plus Amoxicillin

INTERVENTIONS:
Drug: Administration of Metronidazole plus Amoxicillin — Metronidazole plus Amoxicillin after, during and after root planning

SUMMARY:
• Background: Peridontitis is a group of diseases with complex bacterial etiology that affects a large proportion of the Chilean and worldwide population. Its treatment, based on an anti-infective mechanical therapy including scaling and root planning procedures, has been highly effective in numerous short and long term clinical trials. The use of adjunctive systemic antibiotics has shown significant improvements in the initial therapy results of specific periodontal disease types or patient profiles.

The synergic combination of Metronidazole plus amoxicillin has been widely and successfully used for the treatment of aggressive and severe chronic periodontitis, demonstrating additional benefits in clinical and microbiological parameters over scaling and root planning alone. However, and despite its proven efficacy, there is a lack of evidence that evaluates the impact of antimicrobials intake at different times of the mechanical treatment, emphasizing the necessity of a study that compares, simultaneously, the variation of the adjunctive antibiotic effects when they are administered in different moments through the periodontal therapy course.

ELIGIBILITY:
Inclusion Criteria:

* a) age of 35 years old or more, b) at least 3 molars in the mouth, c) at least one site in three of the four quadrants with clinical attachment loss ≥ 3mm; d) at least 4 sites in different teeth with probing depth and clinical attachment level ≥ 6mm and bleeding on probing and at least 14 tooth present in the mouth

Exclusion Criteria:

* a) previous professional root planning; b) systemic/topic antibiotic or antiinflammatory treatment, at least 6 months prior to the initiation of the study; c) immunosuppression or need for antibiotic coverage for routine dental therapy; d) systemic condition that could affect the progression of periodontal disease (diabetes); e) pregnancy or lactation; e) allergy or intolerance to metronidazole or amoxicillin; f) smokers

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
- Mean change in clinical attachment level (CAL) | 12 months

SECONDARY OUTCOMES:
- Mean change in probing pocket depths (PD) | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Odontologia, Santiago, R Metropolitana, Chile